CLINICAL TRIAL: NCT05467839
Title: Evaluation of Efficacy of Microneedling and Topical Methotrexate Versus Microneedling and Topical 5-flourouracil in Treatment of Vitillgo Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Fatma Kassem Ali, Resident of dermatology and venerology at Sohag general hospital, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: soh-med-22-05-10
Record Dates: First submitted 2022-07-04; First posted 2022-07-21 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vitillgo patients (Experimental)
  Interventions: Device: derma pen

INTERVENTIONS:
Device: derma pen — Derma pen is automatic and rechargeable device (vibrating frequency:6500-10000 r/m, vibration speed level 5, model: Ultima A6, company: Dr. Pen and country: Korea). With every case the needle should be replaced. Needle length is adjustable from 0.25mm to 2mm according to the treated areas. The pen is convenient in treating narrow areas such as the nose, around the eye and the mouth. The vibration speed of the pen can be controlled in 5 levels

SUMMARY:
Vitiligo is a depigmenting skin disorder, characterized by the selective loss of melanocytes, which in turn leads to loss of pigment in the affected areas of the skin It considerd as autoimmune disease, associated with genetic and environmental factors together with metabolic, oxidative stress and cell detachment abnormalities The disease affects both genders equally, it can appear at any age, and the average age of onset is somewhat variable in different geographic . with an estimated prevalence of 0.5-2% of the population in both adults and children worldwide 5-Flourouracil is an antimetabolite analogue of the naturally occurring pyrimidine uracil which is metabolised via the same metabolic pathways as uracil Due to its antimitotic activity, topical 5-Flourouracil is a useful therapy for the treatment of many dermatological disorders characterized by a high mitotic rate Clinically, localized hyperpigmentations have been reported during systemic treatment of various cancers by 5-Flourouracil. Usually, these hyperpigmented lesions are located on the normally pigmented extremities (hands and feet) and tongue.

Methotrexate as an antimetabolite and antifolate drug is a time-tested effective treatment extensively used in various autoimmune disorders in low to moderate doses with good efficacy, safety, and tolerability on a long-term basis .

Methotrexate treatment resulted in the decrease of the number of TNF-α-producing T cells, whereas the number of T cells producing IL-10 after polyclonal activation increased, in another study .

ELIGIBILITY:
Inclusion Criteria:

* • Age :main 18 and above years old.

  * Stable vitiligo (each patient has 3separated patches of depigmentation at least).

Exclusion Criteria:• History of keloid formation.

* Patients with systemic diseases (diabetes, bleeding disorders)
* Patients who are receiving chemotherapy or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-31 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
percentage of repigmentation | 6 months
  dermoscopic evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Picardo M, Dell'Anna ML, Ezzedine K, Hamzavi I, Harris JE, Parsad D, Taieb A. Vitiligo. Nat Rev Dis Primers. 2015 Jun 4;1:15011. doi: 10.1038/nrdp.2015.11. PMID 27189851
- [Background] Kruger C, Schallreuter KU. A review of the worldwide prevalence of vitiligo in children/adolescents and adults. Int J Dermatol. 2012 Oct;51(10):1206-12. doi: 10.1111/j.1365-4632.2011.05377.x. Epub 2012 Mar 27. PMID 22458952
- [Background] Feily A. Vitiligo Extent Tensity Index (VETI) score: a new definition, assessment and treatment evaluation criteria in vitiligo. Dermatol Pract Concept. 2014 Oct 31;4(4):81-4. doi: 10.5826/dpc.0404a18. eCollection 2014 Oct. PMID 25396094
- [Background] Ezzedine K, Lim HW, Suzuki T, Katayama I, Hamzavi I, Lan CC, Goh BK, Anbar T, Silva de Castro C, Lee AY, Parsad D, van Geel N, Le Poole IC, Oiso N, Benzekri L, Spritz R, Gauthier Y, Hann SK, Picardo M, Taieb A; Vitiligo Global Issue Consensus Conference Panelists. Revised classification/nomenclature of vitiligo and related issues: the Vitiligo Global Issues Consensus Conference. Pigment Cell Melanoma Res. 2012 May;25(3):E1-13. doi: 10.1111/j.1755-148X.2012.00997.x. PMID 22417114